CLINICAL TRIAL: NCT03273972
Title: INvestigating the Lowest Threshold of Vascular bENefits From LDL Cholesterol Lowering With a PCSK9 mAb InhibiTor (Alirocumab) in healthY Volunteers
Brief Title: INvestigating the Lowest Threshold of Vascular bENefits From LDL Lowering With a PCSK9 InhibiTor in healthY Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant Physician & Clinical Pharmacologist/Associate Lecturer, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: INTENSITY-LOW
Record Dates: First submitted 2017-08-14; First posted 2017-09-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Atherosclerosis; Cardiovascular Diseases
Keywords: Healthy Volunteers; Low Density Lipoprotein Cholesterol (LDL); PCSK9; Alirocumab; Forearm Blood Flow; Arterial Stiffness; Carotid Intima Media Thickness; Inflammation; Endothelial function
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Inflammation | interventions — Pregnancy Tests; Blood Pressure; Heart Rate; Vascular Stiffness; Carotid Intima-Media Thickness; Restraint, Physical; Health Records, Personal; Biomarkers, Pharmacological

STUDY DESIGN:
Intervention Model Description: Randomisation to be performed to a 1:1 ratio.
  Alirocumab treatment arm:
  * V2: Alirocumab (150mg)
  * V3: Alirocumab (150mg) & Atorvastatin (20mg)
  Comparator treatment arm
  * V2: Placebo
  * V3: Placebo & Atorvastatin (20mg)
Who Masked: Participant, Investigator
Masking Description: Independent CRF research nurse to perform the drug administration. CRF nurse will be unblinded whilst the rest of the study team (including the CI/PI) are blinded. This will involve the ACRC nurse bringing the injection in a sealed box to the room, preparing a shield (so the volunteer is blinded), administering the injection (via alirocumab pen or placebo - saline in insulin syringe) and then putting the syringe back in the sealed box and removing the screen. They have to ensure none of the study team are aware of the Rx as well as the patient.
  CRF nurses will also have to collect and store medication in their building. Statin can be stored in a locked cupboard (open label).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alirocumab Treatment Arm (Experimental): V2: Day 1 - Alirocumab 150mg (subcutaneous injection) V3: Day 15 +/- 3 days - Alirocumab 150mg (subcutaneous injection) plus Atorvastatin 20mg (oral) approx. 14 days prescription.
  Interventions: Other: Written Informed Consent; Other: Inclusion/Exclusion check; Other: Full Clinical Chemistry and Haematology Bloods; Other: Serum sample for systemic markers and lipid sub-fractions; Other: Pregnancy Test; Other: 12 Lead ECG; Other: Blood Pressure and Heart Rate; Other: Arterial Stiffness; Other: Central Haemodynamics; Other: Carotid Intima Media Thickness; Other: Forearm blood flow studies; Other: Concomitant medication check; Other: Medication compliance check (Pill count); Other: Physical examination; Other: Medical history; Other: AE/SAE review & reporting; Drug: Dosing
- Comparator Treatment Arm (Other): V2: Day 1 - Placebo (subcutaneous injection) V3: Day 15 +/- 3 days - Placebo (subcutaneous injection) plus Atorvastatin 20mg (oral) approx. 14 days prescription.
  Interventions: Other: Written Informed Consent; Other: Inclusion/Exclusion check; Other: Full Clinical Chemistry and Haematology Bloods; Other: Serum sample for systemic markers and lipid sub-fractions; Other: Pregnancy Test; Other: 12 Lead ECG; Other: Blood Pressure and Heart Rate; Other: Arterial Stiffness; Other: Central Haemodynamics; Other: Carotid Intima Media Thickness; Other: Forearm blood flow studies; Other: Concomitant medication check; Other: Medication compliance check (Pill count); Other: Physical examination; Other: Medical history; Other: AE/SAE review & reporting; Drug: Dosing

INTERVENTIONS:
Other: Written Informed Consent — To be completed prior to conducting any study related procedures
Other: Inclusion/Exclusion check — Eligibility check
Other: Full Clinical Chemistry and Haematology Bloods — Participant required to fast for at least 6-8 hoursprior to visit. (Clear, non-caffeinated fluids are allowed)
Other: Serum sample for systemic markers and lipid sub-fractions — Serum samples may be stored for later analysis.
Other: Pregnancy Test — If applicable for women of child bearing potential
Other: 12 Lead ECG — participant resting supine
Other: Blood Pressure and Heart Rate — Measured in the seated position after 5 minutes rest
Other: Arterial Stiffness — Measure of functional and structural changes which accompanies cardiovascular disease
Other: Central Haemodynamics — Measure of functional and structural changes which accompanies cardiovascular disease
Other: Carotid Intima Media Thickness — Measurements will be repeated three times, and the average of the median values will be recorded
Other: Forearm blood flow studies — Assess and determine vascular function, which can interrogate endothelium dependent and independent mechanisms of nitric oxide bioavailability
Other: Concomitant medication check — Review of medication taken by the participant
Other: Medication compliance check (Pill count) — Ensure prescribed statin has been taken
Other: Physical examination — Check overall health
Other: Medical history — Review of volunteers medial history
Other: AE/SAE review & reporting — Monitor safety from the point of consent
Drug: Dosing — To be performed at the end of the visit following completion all other study visits

SUMMARY:
The INTENSITY-LOW study aims to answer if there are any limits to LDL reduction in relation to benefitting vascular health from a mechanistic viewpoint, and therefore potentially limitations to primary prevention in healthy volunteers by lowering LDL cholesterol using PCSK9 therapies. This research is being carried out because it is unclear what the lowest threshold of LDL cholesterol should be to attain significant reductions in CV risk in healthy individuals. It is also unknown whether there is a true limit of LDL cholesterol below which there is no further improvement in endothelial function in healthy people, and, whether this is associated with a reduction in markers of both systemic and vascular inflammation. This study will hope to provide evidence that the so-called pleiotropic effects of statins are actually mediated by a mechanism of LDL-cholesterol lowering per se and not necessarily a special therapeutic effect of statins.

Defining this may help identify individuals from the general population who may benefit from more aggressive lipid-lowering treatment than standard statin treatment in terms of CV morbidity and mortality.

This study will be conducted in healthy volunteers only, where participants will be randomized to either the Alirocumab arm (which is a therapy designed to lower cholesterol) or comparator arm. Both Alirocumab and comparator arms will be combined with Atorvastatin (another therapy designed to lower cholesterol) at the second dosing visit.

In total, thirty healthy individuals will be recruited to this single centre, randomized, single blind, parallel group, mechanistic physiological study which will be conducted at Cambridge University Hospitals NHS Foundation Trust/University of Cambridge. This study will be open to recruitment for one year and the total study duration for each participant will be approximately 10 weeks. There will be 4 study visits in total with a telephone follow up at the end of the study. Of these visits, two will be dosing visits and the total duration of treatment is approx. 4 weeks.

A series of non-invasive haemodynamic assessments and minimally invasive procedures including blood tests and forearm blood flow measurements will be conducted prior, during and post dosing to determine if there is an improvement of endothelia vascular function (as measured by nitric oxide bioavailability) and reduced systemic inflammation. This study is funded by JP Moulton Charitable Foundation.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy male or female individuals
* Age 18-45 years old inclusive at screening
* Body weight ≥ 45kg and BMI 18 -29.9 kg/m2
* Fasting LDL-C < 4.1 mmol/l, TG <1.7 mmol/l and HDL-C ≥ 1.0 mmol for men and ≥1.3 mmol for women
* Palpable brachial arterial pulse, as per study team assessment
* Not currently eligible for statin therapy according to current treatment criteria

Exclusion Criteria:

* History of established CV disease (Coronary Heart Disease, Cerebrovascular Disease, Peripheral Vascular Disease or Abdominal Aortic Aneurysm)
* Lipid lowering treatment at screening or within 6 weeks before screening
* Pregnancy at any study visit
* Ongoing anticoagulation therapy with warfarin or any of the DOAC/NOAC's
* History of hypersensitivity to any of the study drugs/any known sensitivity to alirocumab or monoclonal antibodies
* History of alcohol or drug abuse or dependence within 6 months of the study at screening
* Current or previous history of regular smoking (defined as 1 pack-year) within the last 10 years.
* History of hypertension or sustained BP ≥140/90 mmHg on repeated measurements at screening
* History of type 1 or 2 diabetes or HbA1c ≥ 48 mmol/mol (6.5%) at screening
* Chronic kidney disease defined as eGFR <60ml/min/1.73m2 at screening
* Biological first-degree relatives who have experienced stroke, TIA, myocardial infarction or peripheral vascular disease (incident event at an age younger than: 55 for male and 65 for female relatives)
* History of autoimmune inflammatory conditions
* Lack of ability to provide informed consent
* TSH >5.0 mu/l at screening
* Clinically significant liver disease on the basis of screening bloods or history
* History of myositis/rhabdomyolysis
* Any concomitant condition that, at the discretion of the investigator, may affect the participants' ability to complete the study or the study results

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Forearm Blood Flow (FBF) - In response to intra-arterial Acetylcholine infusion, comparing Alirocumab to placebo. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography

SECONDARY OUTCOMES:
Forearm Blood Flow in response to intra-arterial Acetylcholine infusion, comparing Alirocumab to statin. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography
Forearm blood flow in response to intra-arterial Acetylcholine infusion, comparing Alirocumab with statin to statin alone. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography
Forearm blood flow in response to intra-arterial Sodium Nitroprusside, comparing Alirocumab to placebo. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography
Forearm blood flow in response to intra-arterial Sodium Nitroprusside, comparing Alirocumab to statin. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography
Forearm blood flow in response to intra-arterial Sodium Nitroprusside, comparing Alirocumab with statin to statin alone. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography
Forearm blood flow in response to intra-arterial L-NMMA infusion, comparing Alirocumab to placebo. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography
Forearm blood flow in response to intra-arterial L-NMMA infusion, comparing Alirocumab to statin. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography
Forearm blood flow in response to intra-arterial L-NMMA infusion, comparing Alirocumab with statin to statin alone. | 4 weeks
  Change in FBF ratio, as measured by absolute & percent change in venous occlusion plethysmography
Total and LDL-cholesterol | 4 weeks
  Correlation of change in responses to Acetylcholine between groups.
Augmentation Index (an indicator of arterial stiffness) | 4 weeks
  Change in Augmentation Index between visits and different treatment regimes.
Pulse Wave Velocity | 4 weeks
  Change in aortic Pulse Wave Velocity between visits and different treatment regimes.
Carotid IMT | 4 weeks
  Change in Carotid IMT between visits and different treatment regimes.
Systemic inflammation | 4 weeks
  Change in lipid profile, hsCRP and other markers of systemic inflammation between visits and different treatment regimes.
Physical examination, vital signs, ECG, laboratory tests and adverse event assessment to determine Safety and tolerability parameters | 4 weeks
  Including physical examination, blood pressure, heart rate, 12-lead electrocardiograms (ECGs), clinical laboratory tests side effects and adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBChB, FRCP, MA, Principal Investigator — Cambridge University Hospitals NHS Trust; Michalis Kostapanos, MD, PhD, FRSPH, Principal Investigator — Cambridge University Hospitals NHS Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only the minimum required participant identifiable information (name and contact details) will be provided to the research team for the purpose of arranging study visits and completing the informed consent process. All delegated research personnel that is responsible to conduct the data/statistical analysis will only analyse data that is anonymised of any patient identifiable data.